CLINICAL TRIAL: NCT05937243
Title: Using Factorial Design to Identify Effective Technological-based Augmentations to Enhance Outcomes From a Smartphone-based Self-help Cognitive Behavior Therapy for Binge Eating
Brief Title: Identifying Effective Technological-based Augmentations to Enhance Outcomes From Self-help Cognitive Behavior Therapy for Binge Eating
Acronym: CONQUER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2205009229
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Binge Eating; Binge-Eating Disorder; Bulimia Nervosa; Bulimia
Keywords: Cognitive behavior therapy; Self-help; Advanced Digital Data Sharing with Coaches; Just-in-time, adaptive interventions; Binge eating; Treatment
MeSH Terms: conditions — Bulimia; Binge-Eating Disorder; Bulimia Nervosa | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: 2*2 factorial design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Base self-help CBT program plus Advanced Digital Data Sharing (ADDS) with Coaches (Experimental): When Advanced DDS with Coaches is turned ON, coaches having a bachelor's degree in health-related fields will have access to a secure web portal called the clinical portal. The portal will also mimic four key behavior change techniques typically employed by an expert clinician including 1) gather data on target behaviors from the base self-help app (i.e., uptake of weekly module, self-monitoring compliance, and skills use), 2) synthesize participants' behavioral data on treatment targets, 3) flag data to indicate behaviors needing improvement and 4) use sophisticated algorithms to generate recommendations for intervening on identified data patterns. Using this information, the coaches will send one weekly email to facilitate improvement in treatment targets over 12 weeks. When Advanced DDS with Coaches is turned OFF, participants' will not have their data shared and will not receive emails from the coaches.
  Interventions: Behavioral: Base self-help CBT program; Behavioral: Advanced Digital Data Sharing (ADDS) with Coaches
- Base self-help CBT program plus Just-in-time, adaptive interventions (JITAIs) (Experimental): When JITAIs are turned ON, the base self-help app will be used to deliver targeted, personalized and automated interventions during algorithm-identified moments when participants could benefit from receiving an intervention for improving two key areas including 1) treatment adherence, and 2) skills utilization based on responses (or lack thereof) in self-help app. When JITAIs are turned OFF, participants will not receive interventions in real-time on the base self-help app.
  Interventions: Behavioral: Base self-help CBT program; Behavioral: Just-in-time, adaptive intervention (JITAIs) system
- Base self-help CBT program plus JITAIs plus Advanced Digital Data Sharing with Coaches (Experimental): When Advanced DDS with Coaches and JITAIs are both ON, participants will receive machine learning-informed interventions. In addition, participants will also receive weekly emails from coaches to provide additional support to improve treatment adherence and skills utilization.
  Interventions: Behavioral: Base self-help CBT program; Behavioral: Just-in-time, adaptive intervention (JITAIs) system; Behavioral: Advanced Digital Data Sharing (ADDS) with Coaches
- Base self-help cognitive behavior therapy (CBT) program (Active Comparator): The self-help app will deliver 12 modules that will be based on Chris Fairburn's "Overcoming Binge Eating" self-help book, the most widely used self-help resource for binge eating. Treatment modules will aim to 1) provide psychoeducation on maintenance factors for binge eating, 2) teach CBT skills designed to interrupt these maintenance factors, and 3) coach participants to set personalized goals each week. Modules will be completed in succession over the course of 12 weeks and a new module will be made open each week. At the end of each weekly module, participants will complete an end-of-the-week survey and report on the frequency of skills use in the past week. In addition, participants will track their eating and eating disorder behaviors using the self-help app.
  Interventions: Behavioral: Base self-help CBT program

INTERVENTIONS:
Behavioral: Base self-help CBT program — The self-help app will deliver 12 modules that will be based on Chris Fairburn's "Overcoming Binge Eating" self-help book, the most widely used self-help resource for binge eating over 12 weeks. Treatment modules will aim to 1) provide psychoeducation on maintenance factors for binge eating, 2) teach CBT skills designed to interrupt these maintenance factors, and 3) coach participant to set personalized goals each week. Modules will be completed in succession over the course of 12-weeks and a new module will be made open each week. In addition, participants will track their eating and eating disorder behaviors using the self-help app.
Behavioral: Just-in-time, adaptive intervention (JITAIs) system — When JITAIs are turned ON, the base self-help app will be used to deliver targeted, personalized and automated interventions during algorithm-identified moments when participants could benefit from receiving an intervention for improving two key areas including 1) treatment adherence, and 2) skills utilization based on responses (or lack thereof) in self-help app. When JITAIs are turned OFF, participants will not receive interventions in real-time on the base self-help app.
  Arms: Base self-help CBT program plus JITAIs plus Advanced Digital Data Sharing with Coaches; Base self-help CBT program plus Just-in-time, adaptive interventions (JITAIs)
Behavioral: Advanced Digital Data Sharing (ADDS) with Coaches — When Advanced DDS with Coaches is turned ON, coaches having a bachelor's degree in health-related fields will have access to a secure web portal called the clinical portal. The portal will also mimic four key behavior change techniques typically employed by an expert clinician including 1) gather data on target behaviors from the base self-help app (i.e., uptake of weekly module, self-monitoring compliance, and skills use), 2) synthesize participants' behavioral data on treatment targets, 3) flag data to indicate behaviors needing improvement and 4) use sophisticated algorithms to generate recommendations for intervening on identified data patterns. Using this information, the coaches will send one weekly email to facilitate improvement in treatment targets over 12 weeks. When Advanced DDS with Coaches is turned OFF, participants' will not have their data shared and will not receive emails from the coaches.
  Arms: Base self-help CBT program plus Advanced Digital Data Sharing (ADDS) with Coaches; Base self-help CBT program plus JITAIs plus Advanced Digital Data Sharing with Coaches

SUMMARY:
The purpose of this study is to test the feasibility, acceptability and efficacy of two technology-based intervention systems (including an Advanced Digital Data Sharing (ADDS) with Coaches or a smartphone-based just-in-time, adaptive interventions (JITAIs) system) for improving treatment adherence, skills utilization and binge eating when used in conjunction with a self-help cognitive behavior therapy [CBT] delivered via a smartphone application [app]). The study is being conducted to test a novel approach to providing evidence-based treatment for binge eating without clinician support in a routine clinical setting.

DETAILED DESCRIPTION:
Self-help cognitive behavior therapies (CBTs) for binge eating are maximally effective when paired with periodic contact with expert clinicians. Clinicians likely improve outcomes because they are trained to utilize specific behavior change techniques for facilitating treatment adherence and skills utilization during self-help CBT programs. Given the limited availability of expert clinicians, it is critical to understand how to enhance outcomes from self-help CBTs without clinician involvement. Technological innovations such as Advanced Digital Data Sharing with Coaches and Just-in-time adaptive interventions (JITAIs) can potentially emulate some of the behavior change techniques used by expert clinicians and improve treatment targets.

The current study will use a 2 x 2 full factorial design in which 76 individuals with bulimia nervosa (BN) or binge eating disorders (BED) are assigned to one of four treatment conditions, i.e., representing each permutation of Advanced DDS with Coaches (Advanced DDS with Coaches ON vs. Advanced DDS with Coaches OFF) and JITAIs (JITAIs ON vs. JITAIs OFF) as an augmentation to self-help CBT program. Self-help CBT will deliver an evidence-based program based on Dr. Chris Fairburn's Overcoming Binge Eating self-help book via a smartphone app without clinician involvement. This app will constitute 12 treatment modules and an electronic self-monitoring form to record eating and eating disorder behaviors for use over 12 weeks without clinician involvement. The primary aims of the study will be to (1) Test target engagement, i.e., that each factor including Advanced DDS with Coach and JITAIs produces greater improvements in treatment adherence and skills utilization, (2) Test the feasibility and acceptability of two intervention factors as adjuncts to self-guided CBT program for binge eating; (3) Test the initial efficacy, i.e., that each factor including Advanced DDS with Coach and JITAIs will produce greater improvements in binge eating frequency at post-treatment, and 3 months follow-up; and (4) Test target validation, i.e., that improvements in treatment adherence and skills utilization will be associated with reductions in binge eating. The exploratory aim will be to quantify the intervention factors' interaction effects, which may be partially additive (because intervention factors overlap and/or there is diminishing return), fully additive, or synergistic (in that intervention factors may partially depend on each other).

ELIGIBILITY:
Inclusion Criteria:

1. Have experienced 12 or more loss of control episodes within the previous 3 months
2. Have a BMI at or above 18.5
3. Are located in the US and willing/able to participate in treatment and assessments
4. Are able to give consent

Exclusion Criteria:

1. Are unable to fluently speak, write and read English
2. Have a BMI below 18.5
3. Are already receiving treatment for an eating disorder
4. Require immediate treatment for medical complications as a result of eating disorder symptoms
5. Have a mental handicap, or are experiencing other severe psychopathology that would limit the participants' ability to comply with the demands of the current study (e.g. severe depression with suicidal intent, active psychotic disorder, severe substance use)
6. Are pregnant or are planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Binge eating frequency | Changes from each assessment time point throughout treatment (3 assessments over 12 weeks) and at a 3 month post-treatment follow-up assessment
  Frequency (number of days and number of instances) of binge eating over the past 28 days assessed by the Eating Disorder Examination
Total number of treatment modules completed | Changes from each assessment time point throughout treatment (3 assessments over 12 weeks) and at a 3 month post-treatment follow-up assessment
  The number of treatment modules completed will be captured from the smartphone application.
Rates of self-monitoring compliance | Changes from each assessment time point throughout treatment (3 assessments over 12 weeks) and at a 3 month post-treatment follow-up assessment
  Number of data entries completed over the course of the treatment will be captured from the smartphone application.
Frequency of skills utilization | Changes from each assessment time point throughout treatment (3 assessments over 12 weeks) and at a 3 month post-treatment follow-up assessment
  Number of times a therapeutic skills was used as indicated by participant on the self-monitored eating records and end-of-the-week surveys.

SECONDARY OUTCOMES:
Severity of Global Eating Pathology | Changes from each assessment time point throughout treatment (3 assessments over 12 weeks) and at a 3 month post-treatment follow-up assessment
  The Eating Disorder Examination is a semi-structured interview that measures eating. pathology. The EDE yields a total eating pathology score that will be used as an outcome variable. Global eating pathology is on a 0-6 point scale with higher scores indicating more significant eating pathology.
Compensatory behavior frequency | Changes from each assessment time point throughout treatment (3 assessments over 12 weeks) and at a 3 month post-treatment follow-up assessment
  Frequency (number of days and number of instances) of compensatory behaviors assessed by the Eating Disorder Examination (EDE)
Acceptability | Changes from each assessment time point throughout treatment after baseline so 2 assessments over 12 weeks (the mid-treatment and post-treatment assessments)
  Perceived usefulness and ease-of-use of the technological components (the smartphone application) will be measured by the Technology Acceptance Model (TAM) Scales. A Feedback Questionnaire will also be used to measure qualitative acceptability of both the technological components of the study and the treatment components.
Acceptability and Feasibility | Changes from each assessment time point throughout treatment after baseline so 2 assessments over 12 weeks (the mid-treatment and post-treatment assessments)
  Assessment of feasibility will include % of eligible patients enrolled, treatment attrition (% of patients that prematurely terminate treatment), and study retention (% of patients that complete all assessment points). Data will also be collected on participants' use of self-help technological features, including time, duration, and frequency of use.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All guidelines for data sharing through the National Database for Clinical Trials Related to Mental Illness (NDCT) and the NIMH Data Archive (NDA) will be duly followed. All de-identified data will be submitted to the NDA at the item level and subject level.
Supporting Information: Study Protocol
Time Frame: Within one year of project completion
Access Criteria: Supporting documentation to allow other researchers to use this data easily and appropriately will be included.

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT05937243/SAP_001.pdf
  • Informed Consent Form (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT05937243/ICF_002.pdf